CLINICAL TRIAL: NCT00586248
Title: A Pilot Study on Pacemaker Interference From Peripheral Nerve Stimulator for
Brief Title: A Pilot Study on Pacemaker Interference From Peripheral Nerve Stimulator for Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Ruei Hsin D Wang,MD, Mayo Clinic Jacksonville
Other Study IDs: 06-002237
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-05

CONDITIONS: Pacemaker, Artificial
Keywords: Peripheral nerve stimulator, cardiac pacemaker

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this prospective pilot study, we proposed to evaluate the effects of left interscalene stimulation on cardiac pacemaker function.

DETAILED DESCRIPTION:
The principle of the nerve stimulation technique consists of using a battery powered peripheral nerve stimulator to generate electrical stimuli through an insulated needle at appropriate anatomical locations. The electrical impulses then trigger depolarization as insulated needle approaches the target nerve bundles. Braun Stimuplex, a common nerve stimulator used for peripheral nerve localization, is currently being used in the United States and other countries. Previous studies have suggested it to be a reliable stimulator for the purpose of peripheral nerve blocks. The operational manual however indicated that this device should not be used in patients with cardiac pacemaker because malfunction of the pacemaker may occur. Literature search on the topic of pacemaker interference from peripheral nerve stimulator showed that there was one case of pacemaker interference caused by activation of a nerve stimulator, resulting in cardiac arrest in a patient with a fixed-rate ventricular pacemaker. Studies and case reports suggest that unipolar electrode seems to be most susceptible to interferences from electrosurgical equipment, TENS unit, spinal cord stimulators. Perhaps this is the reason why the manufacturer of the peripheral nerve stimulator recommends against the use of peripheral nerve stimulator in patients with pacemakers. With the advancements of modern pacemakers technology, it is our experience; interscalene nerve blocks and other peripheral nerve blocks using the nerve stimulator can be performed in patients with pacemakers without notable interferences with pacemaker functions and perhaps the initial recommendation by the peripheral nerve stimulator manufacturer can be modified. In this prospective pilot study, we proposed to evaluate the effects of left interscalene stimulation (most likely scenario to interfere with pacemaker function) by varying the configurations of the pacemaker leads (unipolar vs. bipolar pacer lead configuration) and by varying the positions of the positive electrode of the stimulator.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18, ASA II or III status

Exclusion Criteria:

* Pregnancy, unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3rd degree av block atrial fibrilation chf
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Over sensing of pacemaker during nerve stimulation | during nerve stimulation

SECONDARY OUTCOMES:
Pacemaker mode change during nerve stimulation | during nerve stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Ruei Hsin D Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States

REFERENCES:
- [Background] Skinner HB. Multimodal acute pain management. Am J Orthop (Belle Mead NJ). 2004 May;33(5 Suppl):5-9. PMID 15195936
- [Background] De Andres J, Alonso-Inigo JM, Sala-Blanch X, Reina MA. Nerve stimulation in regional anesthesia: theory and practice. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):153-74. doi: 10.1016/j.bpa.2004.11.002. PMID 15966491
- [Background] Rasmussen MJ, Hayes DL, Vlietstra RE, Thorsteinsson G. Can transcutaneous electrical nerve stimulation be safely used in patients with permanent cardiac pacemakers? Mayo Clin Proc. 1988 May;63(5):443-5. doi: 10.1016/s0025-6196(12)65639-0. PMID 3258950
- [Background] O'Flaherty D, Wardill M, Adams AP. Inadvertent suppression of a fixed rate ventricular pacemaker using a peripheral nerve stimulator. Anaesthesia. 1993 Aug;48(8):687-9. doi: 10.1111/j.1365-2044.1993.tb07181.x. PMID 8214459
- [Background] Kaiser H, Niesel HC, Hans V. [Fundamentals and requirements of peripheral electric nerve stimulation. A contribution to the improvement of safety standards in regional anesthesia]. Reg Anaesth. 1990 Sep;13(7):143-7. German. PMID 2236709